CLINICAL TRIAL: NCT06713434
Title: Pilot, Non-Randomized, Open-Label Study to Determine the Effect of Topical ELK (ELK-003) Eye Drops Applied 6 Times Daily on Ocular Signs and Symptoms in Patients With Junctional and Dystrophic Subtypes of Epidermolysis Bullosa. Estudio Piloto, no Randomizado y Abierto Para Determinar el Efecto de Las Gotas oftalmológicas tópicas ELK Aplicadas 6 Veces al día en Los Signos y síntomas Oculares de Pacientes Con Los Subtipos de la unión y Recesivo distrófico de Epidermólisis Bulosa.
Brief Title: Pilot Study of ELK-003 Eye Drops for Treating Ocular Manifestations of Epidermolysis Bullosa
Acronym: GOTAS-ELK-EB
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fundación DEBRA Chile, Niños Piel de Cristal (Other)
Collaborators: Eliksa Therapeutics, Inc. (Unknown); Centro de la Vision (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-03; 29792/23 (Other: ISP)
Record Dates: First submitted 2024-11-12; First posted 2024-12-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Junctional Epidermolysis Bullosa; Epidermolysis Bullosa (EB); Dystrophic Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa
Keywords: ocular manifestations of EB; corneal abrasion; ELK-003; Debra Chile; Eliksa Therapeutics; Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa, Junctional; Epidermolysis Bullosa; Epidermolysis Bullosa Dystrophica; Corneal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental (Only Arm) (Experimental): In this study, there are two main phases rather than separate arms. During the Observational Phase, no intervention is administered and subjects' natural history of ocular manifestations is documented. In the Treatment Phase, all subjects receive ELK-003 eye drops to assess their effect on ocular sign and symptons. Each subject serves as their own control by comparing outcomes between the Observational and Treatment Phases.
  Interventions: Biological: ELK-003 (Standarized Amniotic Fluid Secretome Eye Drops)

INTERVENTIONS:
Biological: ELK-003 (Standarized Amniotic Fluid Secretome Eye Drops) — ELK-003 eye drops are a standardized amniotic fluid secretome formulation. It contains essential extracellular matrix proteins, such as collagen type VII and laminin-332, which are critical for maintaining corneal integrity in EB patients. In addition, ELK-003 also includes growth factors that stimulate corneal healing and tissue regeneration. This combination of matrix proteins and growth factors aims to enhance corneal surface stability.
  Other Names: ELK-003; Gotas ELK

SUMMARY:
This study consists of two phases: an Observational Phase to evaluate the natural history of ocular manifestations in subjects with Dystrophic and Junctional Epidermolysis Bullosa, followed by a Treatment Phase to assess the effects of ELK-003 eye drops. Each subject will serve as their own control by comparing ocular manifestations documented during the Observational Phase to those recorded during the Treatment Phase.

DETAILED DESCRIPTION:
During this study, subjects will undergo evaluations at three scheduled clinic visits: at enrollment (baseline, time 0), at 4 months, and at the conclusion of the Treatment Phase (6 months post-treatment initiation). Assessments will include OCT imaging, slit lamp examination with photographs, keratograph analysis, visual acuity testing, osmolarity testing, InflammaDry, SPK scoring, Schirmer Test, and opacity scoring. Weekly questionnaires will be completed by subjects to assess symptoms, track corneal abrasions, and evaluate quality of life throughout the study.

If subjects experience symptoms indicative of corneal abrasions, a healthcare provider will conduct a home visit to document the event, using fluorescein staining to confirm and record the corneal abrasion. Corneal abrasion symptoms, frequency, duration, and healing outcomes will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Recessive Dystrophic and Junctional Epidermolysis bullosa
* Frequent history of corneal abrasions (one or more abrasions every 3 months)
* Age: older than 2 years at the time of joining the clinical trial
* Patients and/or parent/legal guardian has given written informed consent in writing

Exclusion Criteria:

* Acute eye infection at time of enrollment
* Patients with severe vision loss (<20/200) or severe corneal opacification.
* Contact lens wear or nocturnal eye ointment
* Hypersensitivity to fluorescein (ocular stain used in slit lamp study)
* History of alcohol abuse or drug addiction
* Patient who reports difficulty to attend the 4 in-person controls
* Patients who are suffering from cancer
* Patients with any medical condition or situation which in the opinion of the investigators could put the patient at risk, or could interfere with the patient's participation in the study
* Pregnant or breastfeeding women (a pregnancy test will be performed using a urine sample for female patients who have had menarche).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety of ELK-003 Eye Drops | 180 days (Treatment Phase)
  The primary outcome is to evaluate the safety and tolerability of ELK-003 eye drops in subjects with EB. Safety assessments will focus on the incidence and severity of drug-related adverse events, including any signs of ocular irritation, monitored throughout the study.

SECONDARY OUTCOMES:
Frequency of Corneal Abrasions (Number of Events) | 180 days (Treatment Phase)
  The secondary outcome is to assess the efficacy of ELK-003 in improving ocular signs and symptoms associated with EB, measuring frequency of corneal abrasions (number of events) over the treatment period.
Days with Corneal Breakdown | 180 days (Treatment Phase)
  The secondary outcome is to assess the efficacy of ELK-003 in improving ocular signs and symptoms associated with EB, measuring days with corneal breakdown over the treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación DEBRA Chile, Niños Piel de Cristal, Santiago, Huechuraba, Chile

IPD SHARING:
Plan to Share IPD: No
We do not plan to share Individual Participant Data with other researchers. However, we plan on publishing the study findings in a peer-reviewed journal.